CLINICAL TRIAL: NCT02918461
Title: A Pilot Study of Emerging From the Haze Evaluating a Trainee-taught Psycho-educational Program to Improve Cancer-related Cognitive Complaints in Gynecologic Cancer Survivors
Brief Title: Emerging From the Haze for Gynecologic Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Arash Asher, MD, Director of Cancer Rehabilitation and Survivorship, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00046105
Record Dates: First submitted 2016-09-21; First posted 2016-09-29 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Gynecologic Neoplasms; Cognition Disorders
MeSH Terms: conditions — Genital Neoplasms, Female; Cognition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emerging from the Haze class (Experimental): A 6-week psycho-educationally-based, cognitive behavioral program to help patients with subjective cognitive complaints after cancer treatment, titled Emerging from the Haze™ (Haze). Each series meets once a week for 2-2.5 hours for 6 weeks.
  Interventions: Behavioral: Emerging from the Haze class

INTERVENTIONS:
Behavioral: Emerging from the Haze class — A 6-week class designed to combat chemotherapy-induced cognitive dysfunction. Patients will report symptoms at 6 months and 1 year after the end of their Haze class.

SUMMARY:
At Cedars-Sinai Medical Center, the investigators have developed a novel curriculum for a 6-week psycho-educationally-based, cognitive behavioral program to help patients with subjective cognitive complaints after cancer treatment, titled Emerging from the Haze™ (Haze). Each series meets once a week for 2-2.5 hours for 6 weeks.

The objective of this study is to quantify the impact of a trainee-taught Emerging from the Haze course on gynecologic cancer survivors' self-report of cognitive changes based on the change of FACT-Cog score.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any stage gynecologic cancer including ovarian, uterine/endometrial, cervical, vulvar, and vaginal cancer
* Treated with chemotherapy solely or in combination with surgery, radiation, and/or hormonal therapy
* Female, age ≥ 18 years.
* FACT-Cog score < 59 on the PCI sub scale
* Eligible after 2 months (60 ±5 days) of completing all their active cancer treatment with the exception of long-term hormonal treatments
* Subjective complaint of cognitive concerns at time of enrollment
* Must be able to understand and communicate proficiently in English
* Ability to understand and the willingness to sign a written informed consent.
* Agree to complete study surveys

Exclusion Criteria:

* Patients who have significant personality disorders or unstable psychiatric disorders (including active major depression, substance abuse, psychosis or bipolar disorder) as assessed by the interviewing clinician
* Patients with known brain metastases, history of brain metastases or radiation to the brain.
* Patients with a history of stroke or other pre-existing neurological condition that may contribute to cognitive dysfunction.
* Non-English speakers
* Receiving treatment for another malignancy other than breast cancer
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, chronic anemia, uncontrolled hypothyroidism, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
The Functional Assessment of Cancer Therapy- Cognition (FACT-Cog) Survey | First day of class (baseline), last day of class (6 weeks), 6 months and 1 year after class
  Measure the change in score from baseline to each of three time points: last day of class (6 weeks), 6 months, and 1 year after class

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) - Cognition and General Concerns Survey | First day of class (baseline), last day of class (6 weeks), 6 months and 1 year after class
  Measure the change in score from baseline to each of three time points: last day of class (6 weeks), 6 months, and 1 year after class
UCLA Loneliness Scale Survey | First day of class (baseline), last day of class (6 weeks), 6 months and 1 year after class
  Measure the change in score from baseline to each of three time points: last day of class (6 weeks), 6 months, and 1 year after class

OTHER OUTCOMES:
Comparison of trainee-taught vs non-trainee taught class | First day of class (baseline), last day of class (6 weeks)
  To compare the impact of a trainee-taught Emerging from the Haze course on gynecologic cancer survivors' self report of cognitive changes based on change of the FACT-Cog compared to the impact of an ongoing non-trainee-taught Emerging from the Haze course on breast cancer survivors' self report of cognitive changes based on the change in FACT-Cog score from first day of class (baseline) to last day of class (6 weeks) in these two groups

CONTACTS AND LOCATIONS:
Overall Officials: Arash Asher, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No